CLINICAL TRIAL: NCT01228383
Title: A Randomized, Single-blind, Active-controlled, Mono-center Phase II Study to Compare the Safety and Neutralizing Activity of Simulated Rabies Post-exposure Prophylaxis With CL184 in Combination With Purified Vero Cell Rabies Vaccine vs. Human Rabies Immune Globulin or Placebo in Combination With Purified Vero Cell Rabies Vaccine vs. CL184 or Placebo in Combination With Human Diploid Cell Rabies Vaccine in Healthy Adult Subjects
Brief Title: Rabies Virus Neutralizing Activity and Safety of CL184, a Monoclonal Antibody Cocktail, in Simulated Rabies Post-Exposure Prophylaxis in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAB-M-A008; U1111-1120-1647 (Other: WHO)
Record Dates: First submitted 2010-10-13; First posted 2010-10-26 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Rabies
Keywords: Monoclonal antibody; Rabies; Post-exposure prophylaxis
MeSH Terms: conditions — Rabies | interventions — Rabies Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- CL184+PVRV (Experimental): CL184 with rabies vaccine (PVRV)
  Interventions: Biological: Rabies virus-specific monoclonal antibodies; Biological: Purified verocell rabies vaccine (PVRV)
- HRIG+PVRV (Active Comparator): HRIG with rabies vaccine
  Interventions: Biological: human polyclonal rabies immune globulin (HRIG); Biological: Purified verocell rabies vaccine (PVRV)
- Placebo+PVRV (Placebo Comparator): Placebo with rabies vaccine (PVRV)
  Interventions: Biological: Placebo; Biological: Purified verocell rabies vaccine (PVRV)
- CL184+HDCV (Experimental): CL184 with rabies vaccine (HDCV)
  Interventions: Biological: Rabies virus-specific monoclonal antibodies; Biological: Human diploid cell vaccine (HDCV)
- Placebo+HDCV (Placebo Comparator): Placebo with rabies vaccine (HDCV)
  Interventions: Biological: Placebo; Biological: Human diploid cell vaccine (HDCV)

INTERVENTIONS:
Biological: Rabies virus-specific monoclonal antibodies — CL184 20 IU/kg intramuscularly on Day 0.
  Other Names: CL184
  Arms: CL184+HDCV; CL184+PVRV
Biological: human polyclonal rabies immune globulin (HRIG) — HRIG 20 IU/kg intramuscularly on Day 0.
  Other Names: Imogam® Rabies-HT
  Arms: HRIG+PVRV
Biological: Placebo — Placebo intramuscularly on Day 0.
  Arms: Placebo+HDCV; Placebo+PVRV
Biological: Human diploid cell vaccine (HDCV) — Rabies vaccine (HDCV) given on Days 0, 3, 7, 14, and 28.
  Other Names: Imovax®
  Arms: CL184+HDCV; Placebo+HDCV
Biological: Purified verocell rabies vaccine (PVRV) — Rabies vaccine (PVRV) given on Days 0, 3, 7, 14, and 28.
  Other Names: Verorab™
  Arms: CL184+PVRV; HRIG+PVRV; Placebo+PVRV

SUMMARY:
Study design:

Single-blind (subject and observer-blinded), active-controlled, randomized [6:2:1:2:1; CL184 + purified vero cell rabies vaccine (PVRV) vs. human rabies immune globulin (HRIG) + PVRV vs. placebo + PVRV vs. CL184 + human diploid cell vaccine (HDCV) vs. placebo + HDCV], mono-center study

Study objectives:

Primary: To evaluate the safety of CL184 in combination with PVRV in healthy adult subjects.

Secondary: To evaluate the safety of HRIG or placebo in combination with PVRV and to evaluate the safety of CL184 or placebo in combination with HDCV in healthy adult subjects. To evaluate the rabies virus neutralizing activity (RVNA) after administration of CL184 or placebo in combination with PVRV, of HRIG in combination with PVRV, and of CL184 or placebo in combination with HDCV in healthy adult subjects. To evaluate the pharmacokinetics of the monoclonal antibodies (mAbs).

DETAILED DESCRIPTION:
This study was designed to explore and obtain further safety and RVNA data on CL184 in comparison to HRIG and placebo as part of a classical post-exposure prophylaxis (PEP) regimen. This regimen will be applied as simulated PEP regimen to healthy subjects (i.e. in a pre-exposure setting) in this study. A comparison with placebo combined with each rabies vaccine was included to differentiate between the contribution of immune globulin and vaccine and to investigate potential interactions between immune globulin and vaccine. RVNA provided by CL184 or HRIG, as well as vaccination response will be checked regularly during the study and booster doses can be applied after the study, if necessary. In addition pharmacokinetic data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged ≥18 to ≤55 years
* Subjects free of obvious health-problems or with stable conditions or medications
* Body mass index between ≥18 to ≤30 kg/m2
* Abstinence from sexual intercourse or use of adequate contraception from the date of screening up to Day 90
* Male subjects must agree that they will not donate sperm from the first check-in until Day 90
* Subject signed written informed consent

Exclusion Criteria:

* Prior history of active or passive rabies immunization
* Clinically significant acute illness or infection including fever (≥38 °C) within 2 weeks before first dosing
* History and/or family history of clinically significant immunodeficiency or auto-immune disease
* Planned immunization with live vaccines during the coming 3 months after first dosing
* Chronic (longer than 14 days) administration of immunosuppressants or other immune-modifying drugs within 6 months before the first dose of investigational medicinal product

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2011-12; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety | 90 days
  Assessed by recording unsolicited adverse events, solicited local and systemic adverse events, and pain at the injection site (assessed on a Visual Analog Scale from Day 0 to Day 3); routine safety laboratory assessed on Days -1, 1, 3, 7, 42, and 90; ECG and vital signs assessed on Days -1, 7, and 90.

SECONDARY OUTCOMES:
Rabies virus neutralizing activity | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: G Nagashayana, MD, Principal Investigator — Lotus Labs Pvt. Ltd, Bangalore, India
Locations (1):
- Lotus House, Vasanth Nagar, Bangalore, Karnataka, India